CLINICAL TRIAL: NCT03070119
Title: An Extension Study to Assess the Long-Term Safety, Tolerability, Pharmacokinetics, and Effect on Disease Progression of BIIB067 Administered to Previously Treated Adults With Amyotrophic Lateral Sclerosis Caused by Superoxide Dismutase 1 Mutation
Brief Title: Long-Term Evaluation of BIIB067 (Tofersen)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 233AS102; 2016-003225-41 (EudraCT Number)
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: ALS Caused by Superoxide Dismutase 1 (SOD1) Mutation
MeSH Terms: interventions — tofersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIIB067 (Experimental): Participants who have completed Parts A, B, or C of study 233AS101 will be placed in this arm.
  Interventions: Drug: Tofersen

INTERVENTIONS:
Drug: Tofersen — Participants will receive a loading dose regimen followed by maintenance dosing.
  Other Names: BIIB067; QALSODY

SUMMARY:
The primary objective of the study is to evaluate the long-term safety and tolerability of BIIB067 (tofersen) in participants with amyotrophic lateral sclerosis (ALS) and confirmed superoxide dismutase 1 (SOD1) mutation. The secondary objectives are to evaluate the pharmacokinetic (PK), pharmacodynamic (PD), biomarker effects, and efficacy of BIIB067 administered to participants with ALS and a confirmed SOD1 mutation.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have diagnosis of superoxide dismutase 1-amyotrophic lateral sclerosis (SOD1-ALS), and must have completed the End of Study Visit for either Parts A, B, or C of Study 233AS101 (NCT02623699) (i.e., were not withdrawn).
* If taking riluzole, participant must be receiving a stable dose for ≥30 days prior to Day 1.
* If taking edaravone, participant must have initiated edaravone ≥60 days (2 treatment cycles) prior to Day 1. Edaravone may not be administered on dosing days during this study.
* Medically able to undergo the study procedures, and to adhere to the visit schedule at the time of study entry, as determined by the Investigator.
* For female participants of childbearing potential must agree to practice effective contraception during the study and be willing and able to continue contraception for 5 months after their last dose of study treatment.
* Participants from Study 233AS101 Parts A and B must have a washout ≥16 weeks between the last dose of study treatment received in Study 233AS101 and the first dose of BIIB067 received in the current Study 233AS102.

Key Exclusion Criteria:

* History of allergies to a broad range of anesthetics.
* Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that is not managed optimally and could place a participant at an increased risk for bleeding during or after a Lumbar Puncture (LP) procedure. These risks could include, but are not limited to, anatomical factors at or near the LP site (e.g., vascular abnormalities, neoplasms, or other abnormalities) and underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., hemophilia, Von Willebrand's disease, liver disease).
* Presence of an implanted shunt for the drainage of CSF or an implanted central nervous system (CNS) catheter.
* Prior or current treatment with small interfering ribonucleic acid (RNA), stem cell therapy, or gene therapy.
* Treatment with another investigational drug, biological agent (excluding BIIB067), or device within 1 month or 5 half-lives of study agent, whichever is longer.
* Current or anticipated need, in the opinion of the Investigator, of a diaphragm pacing system (DPS) during the study period.
* Current or recent (within 1 month) use, or anticipated need, in the opinion of the Investigator, of copper (II) (diacetyl-bis(N4-methylthiosemicarbazone)) or pyrimethamine.
* Female participants who are pregnant or currently breastfeeding.
* Current enrollment in any other interventional study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (30):
- United States (16):
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, San Francisco, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Knoxville, Tennessee
- Research Site, Leuven, Belgium
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Bispebjerg Hospital, Copenhagen, Denmark
- Research Site, Clermont-Ferrand, Puy De Dome, France
- Research Site, Ulm, Baden-Wurttemberg, Germany
- Research Site, Torino, Italy
- Japan (4):
  - Research Site, Bunkyō City
  - Research Site, Kagoshima
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
- Research Site, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Miller TM, Cudkowicz ME, Shaw PJ, Genge A, Sobue G, Bucelli RC, Chio A, Van Damme P, Ludolph AC, Glass JD, Andrews JA, Babu S, Benatar M, McDermott CJ, Salachas F, Bruneteau G, Al-Chalabi A, Amorin M, Nestorov I, Graham D, Lin L, Sun P, McNeill M, Malek S, Inra J, Garafalo S, Fradette S; VALOR and OLE Working Group. Long-Term Tofersen in SOD1 Amyotrophic Lateral Sclerosis. JAMA Neurol. 2026 Feb 1;83(2):115-125. doi: 10.1001/jamaneurol.2025.4946. PMID 41661214
- [Derived] Miller TM, Cudkowicz ME, Genge A, Shaw PJ, Sobue G, Bucelli RC, Chio A, Van Damme P, Ludolph AC, Glass JD, Andrews JA, Babu S, Benatar M, McDermott CJ, Cochrane T, Chary S, Chew S, Zhu H, Wu F, Nestorov I, Graham D, Sun P, McNeill M, Fanning L, Ferguson TA, Fradette S; VALOR and OLE Working Group. Trial of Antisense Oligonucleotide Tofersen for SOD1 ALS. N Engl J Med. 2022 Sep 22;387(12):1099-1110. doi: 10.1056/NEJMoa2204705. PMID 36129998

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and took part at the investigative sites in Belgium, Canada, France, Germany, Italy, Japan, Denmark, the United Kingdom, and the United States from 08 Mar 2017 to 12 Aug 2024.
Pre-assignment Details: A total of 139 participants were randomized in the study, of which 95 participants rolled over from Part C and 44 participants rolled over from Parts A and B of the parent study 233AS101 (NCT02623699).
Groups:
- 233AS101: Part C (Prior Placebo): Participants who were randomized to placebo in Part C of the parent study 233AS101 received 3 loading doses of BIIB067, 100 milligrams (mg), once every 2 weeks (Q2W), on Days 1, 15, and 29 by intrathecal (IT) bolus injection in this study followed by up to 90 maintenance doses of BIIB067, every 4 weeks (Q4W), until the last enrolled participant had their Week 152 maintenance dose visit.
- 233AS101: Part C (Prior BIIB067 100 mg): Participants who were randomized to BIIB067 100 mg in Part C of the parent study 233AS101 received 2 loading doses of BIIB067, 100 mg, on Days 1 and 29, and one dose of BIIB067-matched placebo on Day 15 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067,Q4W, until the last enrolled participant had their Week 152 maintenance dose visit.
- 233AS101: Part A and B (All Doses): Participants who were randomized to BIIB067 or placebo in Part A (at doses 10 mg, 20 mg, 40 mg and 60 mg) or Part B (at doses 20 mg, 40 mg, 60 mg and 100 mg) of the parent study 233AS101 received 3 loading doses of BIIB067, 20 mg, 40 mg, 60 mg, or 100 mg, eventually escalated to 100 mg, 2 weeks apart, and up to 90 maintenance doses, Q4W, by IT bolus injection until the last enrolled participant had their Week 152 maintenance dose visit in this study.
Period: Overall Study
Arm/Group | 233AS101: Part C (Prior Placebo) | 233AS101: Part C (Prior BIIB067 100 mg) | 233AS101: Part A and B (All Doses)
Started | 32 | 63 | 44
Completed | 12 | 34 | 26
Not Completed | 20 | 29 | 18
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Consent Withdrawn | 6 | 5 | 3
Not completed — Investigator Decision | 0 | 0 | 1
Not completed — Death | 7 | 14 | 5
Not completed — Disease Progression | 5 | 7 | 7
Not completed — Reason not Specified | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who were enrolled and received at least one dose of study treatment in 233AS102.
Groups:
- 233AS101: Part C (Prior Placebo): Participants who were randomized to placebo in Part C of the parent study 233AS101 received 3 loading doses of BIIB067, 100mg, Q2W, on Days 1, 15, and 29 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067, Q4W, until the last enrolled participant had their Week 152 maintenance dose visit.
- Total: Total of all reporting groups
Arm/Group | 233AS101: Part C (Prior Placebo) | 233AS101: Part C (Prior BIIB067 100 mg) | 233AS101: Part A and B (All Doses) | Total
Number analyzed (Participants) | 32 | 63 | 44 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (11.00) | 48.1 (11.80) | 49.8 (11.04) | 49.7 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 24 | 19 | 58
  Male | 17 | 39 | 25 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 4
  Not Hispanic or Latino | 25 | 40 | 26 | 91
  Unknown or Not Reported | 6 | 20 | 18 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 4 | 4 | 1 | 9
  Race: Black or African American | 0 | 1 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Race: White | 22 | 37 | 23 | 82
  Race: Not Reported | 6 | 20 | 18 | 44
  Race: Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious AEs (TESAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, life-threatening event, requires inpatient hospitalization, significant disability/incapacity or congenital anomaly. TEAEs were defined as any AEs or SAE with an onset date and time that was on or after the first dose of study drug, or any pre-existing condition that worsened in severity after the first dose of study drug.
Time Frame: From first dose of the study drug in the current study up to end of follow-up period (up to Week 364)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 233AS101: Part C (Prior Placebo) | 233AS101: Part C (Prior BIIB067 100 mg) | 233AS101: Part A and B (All Doses)
Number analyzed (Participants) | 32 | 63 | 44
Participants
  TEAEs | 31 | 63 | 43
  TESAEs | 16 | 33 | 22

2. Secondary Outcome: Plasma Concentration of BIIB067
Time Frame: Week 4
Population: As planned, plasma concentration of BIIB067 was summarized for 233AS101 Part C participants only. Pharmacokinetic (PK) population included all participants who received at least 1 dose of study treatment & had at least 1 post-dosing PK concentration measurement in current study. 'Overall number of participants analyzed' indicates the number of participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | 233AS101: Part C (Prior Placebo) | 233AS101: Part C (Prior BIIB067 100 mg)
Number analyzed (Participants) | 28 | 60
nanograms per milliliter (ng/mL) | 1.22 (0.118) | 2.05 (0.516)

3. Secondary Outcome: Concentration of BIIB067 in Cerebrospinal Fluid (CSF)
Time Frame: Week 4
Population: As planned, concentration of BIIB067 in CSF was summarized for 233AS101 Part C participants only. PK population included all participants who received at least 1 dose of study treatment & had at least 1 post-dosing PK concentration measurement in current study. 'Overall number of participants analyzed' indicates the number of participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 233AS101: Part C (Prior Placebo) | 233AS101: Part C (Prior BIIB067 100 mg)
Number analyzed (Participants) | 25 | 47
ng/mL | 19.35 (2.829) | 9.18 (0.711)

4. Secondary Outcome: 233AS101 and 233AS102 Integrated Summary of Efficacy (ISE): Total CSF Superoxide Dismutase 1 (SOD1) Protein Ratio to Baseline
Description: This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on the data collected from both 233AS101 and 233AS102 studies. This is reported as a part of the final integrated analyses. Baseline is defined as the Day 1 of 233AS101 Part C. Data has been reported for Weeks 52, 104 and 148 from the 233AS101 Part C baseline.
Time Frame: Baseline, Weeks 52, 104 and 148
Population: Integrated analysis was performed on overall ITT population which included all Part C participants of 233AS101 and participants who rolled over from 233AS101 Part C into 233AS102. 'Overall number of participants analyzed' exceeds the total number of participants who started study 233AS102 as it indicates participants who were randomized in the Part C 233AS101 study. Number analyzed 'n' indicates the number of participants evaluable for this outcome measure at specified time point.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg: Participants who were randomized to placebo in Part C of the parent study 233AS101 received 3 loading doses of BIIB067, 100 mg, Q2W, on Days 1, 15, and 29 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067, Q4W, until the last enrolled participant had their Week 152 maintenance dose visit.
- 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg: Participants who were randomized to BIIB067 100 mg in Part C of the parent study 233AS101 received 2 loading doses of BIIB067, 100 mg, on Days 1 and 29, and one dose of BIIB067-matched placebo on Day 15 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067,Q4W, until the last enrolled participant had their Week 152 maintenance dose visit.
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
ratio
  Week 52: number analyzed (Participants) | 25 | 52
  Week 52 | 0.78 [0.64 to 0.96] | 0.67 [0.57 to 0.79]
  Week 104: number analyzed (Participants) | 17 | 44
  Week 104 | 0.81 [0.67 to 0.97] | 0.74 [0.65 to 0.84]
  Week 148: number analyzed (Participants) | 11 | 41
  Week 148 | 0.75 [0.61 to 0.92] | 0.79 [0.69 to 0.91]
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 52 - The analysis was based on an analysis of covariance (ANCOVA) model with natural log transformed data. The model included covariates for the corresponding baseline value i.e. log value, and use of riluzole or edaravone. Multiple imputation (MI) including treatment group, use of riluzole or edaravone, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; Least square (LS) geometric mean ratio = 0.86, 95% CI 2-sided [0.69 to 1.08]
Statistical Analysis 2: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 104 - The analysis was based on an ANCOVA model with natural log transformed data. The model included covariates for the corresponding baseline value i.e. log value, and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.3711, ANCOVA; ANCOVA model using MI; LS geometric mean ratio = 0.91, 95% CI 2-sided [0.75 to 1.11]
Statistical Analysis 3: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 148 - The analysis was based on an ANCOVA model with natural log transformed data. The model included covariates for the corresponding baseline value i.e. log value, and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.6344, ANCOVA; ANCOVA model using MI; LS geometric mean ratio = 1.06, 95% CI 2-sided [0.84 to 1.34]

5. Secondary Outcome: 233AS101 and 233AS102 ISE: Neurofilament Light Chain (NfL) Plasma Concentration Ratio to Baseline
Description: as for outcome 4
Time Frame: Baseline, Weeks 52, 104 and 148
Population: as for outcome 4
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg: Participants who were randomized to BIIB067 100 mg in Part C of the parent study 233AS101 received 2 loading doses of BIIB067, 100 mg, on Days 1 and 29, and one dose of BIIB067-matched placebo on Day 15 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067, Q4W, until the last enrolled participant had their Week 152 maintenance dose visit.
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
ratio
  Week 52: number analyzed (Participants) | 23 | 50
  Week 52 | 0.62 [0.49 to 0.78] | 0.50 [0.42 to 0.60]
  Week 104: number analyzed (Participants) | 18 | 42
  Week 104 | 0.41 [0.30 to 0.55] | 0.33 [0.27 to 0.42]
  Week 148: number analyzed (Participants) | 11 | 41
  Week 148 | 0.36 [0.25 to 0.53] | 0.33 [0.26 to 0.43]
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 52 - The analysis was based on an ANCOVA model with natural log transformed data. The model included covariates for the corresponding baseline value i.e. log value, and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; LS geometric mean ratio = 0.8, 95% CI 2-sided [0.63 to 1.03]
Statistical Analysis 2: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.2306, ANCOVA; ANCOVA model using MI; LS geometric mean ratio = 0.83, 95% CI 2-sided [0.60 to 1.13]
Statistical Analysis 3: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.6730, ANCOVA; ANCOVA model using MI; LS geometric mean ratio = 0.92, 95% CI 2-sided [0.61 to 1.38]

6. Secondary Outcome: 233AS101 and 233AS102 ISE: Change From Baseline in Total Amyotropic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) Score
Description: The ALSFRS-R measures 4 functional domains, including respiratory, bulbar function, gross motor skills, and fine motor skills. There are 12 questions, each scored from 0 (no function) to 4 (full function). The ALSFRS-R total score was calculated as the sum of the 4 functional domain scores, ranging from 0 to 48, where higher scores representing better function. Negative change from baseline indicates disease progression. This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on the data collected from both 233AS101 and 233AS102 studies. This is reported as a part of the final integrated analyses. Baseline is defined as the Day 1 of 233AS101 Part C. Data has been reported for Weeks 52, 104 and 148 from the 233AS101 Part C baseline.
Time Frame: Baseline, Weeks 52, 104 and 148
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
score on a scale
  Week 52: number analyzed (Participants) | 28 | 57
  Week 52 | -9.5 (1.46) | -5.9 (1.16)
  Week 104: number analyzed (Participants) | 20 | 49
  Week 104 | -13.1 (2.12) | -9.4 (1.69)
  Week 148: number analyzed (Participants) | 13 | 46
  Week 148 | -13.5 (2.28) | -9.9 (1.77)
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 52 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline ALSFRS-R total score, and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; Least square (LS) mean difference = 3.6, 95% CI 2-sided [0.5 to 6.7], Standard Error of Mean 1.58
Statistical Analysis 2: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 104 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline ALSFRS-R total score, and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.1054, ANCOVA; ANCOVA model using MI; LS mean difference = 3.7, 95% CI 2-sided [-0.8 to 8.2], Standard Error of Mean 2.28
Statistical Analysis 3: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 148 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline ALSFRS-R total score, and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.1432, ANCOVA; ANCOVA model using MI; LS mean difference = 3.6, 95% CI 2-sided [-1.2 to 8.4], Standard Error of Mean 2.46

7. Secondary Outcome: 233AS101 and 233AS102 ISE: Change From Baseline in Percent Predicted Slow Vital Capacity (SVC)
Description: Vital capacity was measured by means of an SVC test, administered in the upright position. Upright SVC was determined by performing 3 to 5 measures, in accordance with criteria established by the American Thoracic Society and the European Respiratory Society. The percent predicted SVC was calculated as [observed SVC divided by predicted SVC]*100%. The predicted SVC was adjusted by sex, age, height, which was programmed into and performed by the equipment used. Negative change from baseline indicated worsening of respiratory capacity. This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on the data collected from both 233AS101 and 233AS102 studies. This is reported as a part of the final integrated analyses. Baseline is defined as the Day 1 of 233AS101 Part C. Data has been reported for Weeks 52, 104 and 148 from the 233AS101 Part C baseline.
Time Frame: Baseline, Weeks 52, 104 and 148
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted volume
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
percentage of predicted volume
  Week 52: number analyzed (Participants) | 20 | 38
  Week 52 | -18.7 (3.70) | -10.6 (2.99)
  Week 104: number analyzed (Participants) | 10 | 31
  Week 104 | -23.7 (5.90) | -14.4 (4.46)
  Week 148: number analyzed (Participants) | 10 | 32
  Week 148 | -18.1 (5.74) | -13.8 (4.07)
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 52 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline percent predicted SVC and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; LS mean difference = 8.1, 95% CI 2-sided [0.3 to 15.9], Standard Error of Mean 3.99
Statistical Analysis 2: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 104 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline percent predicted SVC and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.0963, ANCOVA; ANCOVA model using MI; LS mean difference = 9.3, 95% CI 2-sided [-1.7 to 20.4], Standard Error of Mean 5.6
Statistical Analysis 3: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 148 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline percent predicted SVC and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.4388, ANCOVA; ANCOVA model using MI; LS mean difference = 4.3, 95% CI 2-sided [-6.6 to 15.2], Standard Error of Mean 5.56

8. Secondary Outcome: 233AS101 and 233AS102 ISE: Change From Baseline in Handheld Dynamometry (HHD) Overall Megascore
Description: Quantitative muscle strength was evaluated using the HHD Megascore, which tests isometric strength of multiple muscles using standard participant positioning. Approximately 8 muscle groups were examined (per each side) in both upper and lower extremities. The muscle strength values were normalized to Z scores as (post-baseline measurements - mean)/SD and averaged to provide HHD overall megascore. The overall megascore was created by averaging all eight bilateral measurement Z scores, if no more than 10 (≤ 10) measures are missing. A negative change from baseline indicated decreased muscle strength. This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on the data collected from both 233AS101 and 233AS102 studies. This is reported as a part of the final integrated analyses. Baseline is defined as the Day 1 of 233AS101 Part C. Data has been reported for Weeks 52, 104 and 148 from the 233AS101 Part C baseline.
Time Frame: Baseline, Weeks 52, 104 and 148
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
score on a scale
  Week 52: number analyzed (Participants) | 25 | 42
  Week 52 | -0.41 (0.101) | -0.15 (0.079)
  Week 104: number analyzed (Participants) | 10 | 32
  Week 104 | -0.56 (0.154) | -0.42 (0.112)
  Week 148: number analyzed (Participants) | 10 | 36
  Week 148 | -0.43 (0.089) | -0.38 (0.062)
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 52 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline HHD overall megascore and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; LS mean difference = 0.26, 95% CI 2-sided [0.051 to 0.477], Standard Error of Mean 0.109
Statistical Analysis 2: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 104 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline HHD overall megascore and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.3207, ANCOVA; ANCOVA model using MI; LS mean difference = 0.14, 95% CI 2-sided [-0.141 to 0.430], Standard Error of Mean 0.145
Statistical Analysis 3: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Week 148 - The analysis was based on an ANCOVA model that included treatment as a fixed effect and adjusted for the following covariates: baseline plasma NfL, baseline HHD overall megascore and use of riluzole or edaravone. Multiple imputation including treatment group, use of riluzole or edaravone, baseline NfL, and the relevant baseline and postbaseline values for the endpoint was used for missing data; Test type: Superiority; p = 0.5452, ANCOVA; ANCOVA model using MI; LS mean difference = 0.06, 95% CI 2-sided [-0.124 to 0.234], Standard Error of Mean 0.091

9. Secondary Outcome: 233AS101 and 233AS102 ISE: Change From Baseline in Individual Muscle Strength Assessed by HHD
Description: Individual muscle strength was evaluated using handheld dynamometer which tests the isometric strength of multiple muscles using standard participant positioning. Eight muscle groups were examined (per each side) in both upper and lower extremities. Negative change from baseline=decreased muscle strength. The analyses was based on observed data. This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on data collected from both 233AS101 & 233AS102 studies. This is reported as a part of final integrated analyses.
Time Frame: Baseline, Weeks 52, 104 and 148
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
kilogram (kg)
  Left Shoulder Flexion: Week 52: number analyzed (Participants) | 25 | 41
  Left Shoulder Flexion: Week 52 | -3.42 (6.671) | -0.51 (8.484)
  Left Shoulder Flexion: Week 104: number analyzed (Participants) | 10 | 32
  Left Shoulder Flexion: Week 104 | 0.17 (5.714) | -4.16 (14.329)
  Left Shoulder Flexion: Week 148: number analyzed (Participants) | 10 | 36
  Left Shoulder Flexion: Week 148 | -2.48 (5.075) | -4.12 (8.543)
  Left Elbow Flexion: Week 52: number analyzed (Participants) | 25 | 42
  Left Elbow Flexion: Week 52 | -3.89 (6.747) | -0.24 (8.031)
  Left Elbow Flexion: Week 104: number analyzed (Participants) | 10 | 32
  Left Elbow Flexion: Week 104 | -1.26 (7.361) | -3.12 (13.334)
  Left Elbow Flexion: Week 148: number analyzed (Participants) | 10 | 36
  Left Elbow Flexion: Week 148 | 0.65 (4.560) | -3.33 (8.753)
  Left Wrist Extension: Week 52: number analyzed (Participants) | 25 | 41
  Left Wrist Extension: Week 52 | -3.66 (4.775) | -0.41 (7.170)
  Left Wrist Extension: Week 104: number analyzed (Participants) | 10 | 32
  Left Wrist Extension: Week 104 | -0.86 (5.279) | -1.74 (8.517)
  Left Wrist Extension: Week 148: number analyzed (Participants) | 10 | 36
  Left Wrist Extension: Week 148 | 0.95 (5.242) | -2.49 (6.086)
  Left Abduction Index Finger (First Dorsal Interosseous): Week 52: number analyzed (Participants) | 25 | 42
  Left Abduction Index Finger (First Dorsal Interosseous): Week 52 | -0.96 (1.450) | -0.93 (4.448)
  Left Abduction Index Finger (First Dorsal Interosseous): Week 104: number analyzed (Participants) | 10 | 32
  Left Abduction Index Finger (First Dorsal Interosseous): Week 104 | -0.63 (1.266) | -0.62 (2.279)
  Left Abduction Index Finger (First Dorsal Interosseous): Week 148: number analyzed (Participants) | 10 | 36
  Left Abduction Index Finger (First Dorsal Interosseous): Week 148 | -0.41 (1.604) | -1.28 (4.913)
  Left Abduction Thumb (Abductor Pollicus Brevis): Week 52: number analyzed (Participants) | 25 | 41
  Left Abduction Thumb (Abductor Pollicus Brevis): Week 52 | -1.15 (1.486) | -0.70 (2.497)
  Left Abduction Thumb (Abductor Pollicus Brevis): Week 104: number analyzed (Participants) | 10 | 32
  Left Abduction Thumb (Abductor Pollicus Brevis): Week 104 | -0.69 (1.089) | -0.19 (2.382)
  Left Abduction Thumb (Abductor Pollicus Brevis): Week 148: number analyzed (Participants) | 10 | 36
  Left Abduction Thumb (Abductor Pollicus Brevis): Week 148 | -1.10 (2.324) | -0.78 (3.049)
  Left Abduction 5th Digit (Abductor Digiti Minimi): Week 52: number analyzed (Participants) | 25 | 41
  Left Abduction 5th Digit (Abductor Digiti Minimi): Week 52 | -0.66 (1.208) | -0.49 (2.296)
  Left Abduction 5th Digit (Abductor Digiti Minimi): Week 104: number analyzed (Participants) | 10 | 31
  Left Abduction 5th Digit (Abductor Digiti Minimi): Week 104 | -0.47 (1.226) | -0.50 (1.999)
  Left Abduction 5th Digit (Abductor Digiti Minimi): Week 148: number analyzed (Participants) | 10 | 36
  Left Abduction 5th Digit (Abductor Digiti Minimi): Week 148 | -0.43 (1.496) | -0.66 (2.394)
  Left Knee Extension: Week 52: number analyzed (Participants) | 25 | 42
  Left Knee Extension: Week 52 | -4.94 (8.015) | 1.80 (10.744)
  Left Knee Extension: Week 104: number analyzed (Participants) | 10 | 32
  Left Knee Extension: Week 104 | -2.41 (6.545) | -1.54 (13.222)
  Left Knee Extension: Week 148: number analyzed (Participants) | 10 | 35
  Left Knee Extension: Week 148 | -2.48 (7.339) | -2.01 (9.711)
  Left Ankle Dorsiflexion: Week 52: number analyzed (Participants) | 25 | 42
  Left Ankle Dorsiflexion: Week 52 | -2.82 (7.560) | 0.72 (7.701)
  Left Ankle Dorsiflexion: Week 104: number analyzed (Participants) | 10 | 31
  Left Ankle Dorsiflexion: Week 104 | -5.47 (3.590) | -4.20 (11.516)
  Left Ankle Dorsiflexion: Week 148: number analyzed (Participants) | 10 | 35
  Left Ankle Dorsiflexion: Week 148 | -5.43 (5.303) | -2.33 (9.533)
  Right Shoulder Flexion: Week 52: number analyzed (Participants) | 25 | 41
  Right Shoulder Flexion: Week 52 | -4.74 (5.494) | -0.96 (5.728)
  Right Shoulder Flexion: Week 104: number analyzed (Participants) | 10 | 32
  Right Shoulder Flexion: Week 104 | -2.72 (4.638) | -2.81 (9.304)
  Right Shoulder Flexion: Week 148: number analyzed (Participants) | 10 | 36
  Right Shoulder Flexion: Week 148 | -3.02 (5.066) | -3.18 (8.139)
  Right Elbow Flexion: Week 52: number analyzed (Participants) | 25 | 41
  Right Elbow Flexion: Week 52 | -4.03 (5.663) | -1.20 (7.015)
  Right Elbow Flexion: Week 104: number analyzed (Participants) | 10 | 31
  Right Elbow Flexion: Week 104 | -1.32 (6.289) | -3.04 (9.717)
  Right Elbow Flexion: Week 148: number analyzed (Participants) | 10 | 35
  Right Elbow Flexion: Week 148 | 0.49 (3.407) | -3.28 (8.704)
  Right Wrist Extension: Week 52: number analyzed (Participants) | 25 | 42
  Right Wrist Extension: Week 52 | -3.82 (5.892) | -0.63 (4.870)
  Right Wrist Extension: Week 104: number analyzed (Participants) | 10 | 32
  Right Wrist Extension: Week 104 | -0.76 (4.086) | -1.65 (6.267)
  Right Wrist Extension: Week 148: number analyzed (Participants) | 10 | 36
  Right Wrist Extension: Week 148 | 0.09 (5.096) | -1.89 (5.033)
  Right Abduction Index Finger (First Dorsal Interosseous): Week 52: number analyzed (Participants) | 25 | 42
  Right Abduction Index Finger (First Dorsal Interosseous): Week 52 | -0.86 (1.381) | -0.36 (1.405)
  Right Abduction Index Finger (First Dorsal Interosseous): Week 104: number analyzed (Participants) | 10 | 31
  Right Abduction Index Finger (First Dorsal Interosseous): Week 104 | -0.38 (1.057) | -0.45 (1.569)
  Right Abduction Index Finger (First Dorsal Interosseous): Week 148: number analyzed (Participants) | 10 | 36
  Right Abduction Index Finger (First Dorsal Interosseous): Week 148 | -0.23 (1.545) | -0.46 (1.193)
  Right Abduction Thumb (Abductor Pollicus Brevis): Week 52: number analyzed (Participants) | 25 | 41
  Right Abduction Thumb (Abductor Pollicus Brevis): Week 52 | -0.98 (1.425) | -1.24 (4.595)
  Right Abduction Thumb (Abductor Pollicus Brevis): Week 104: number analyzed (Participants) | 10 | 32
  Right Abduction Thumb (Abductor Pollicus Brevis): Week 104 | -0.31 (0.947) | -0.24 (2.016)
  Right Abduction Thumb (Abductor Pollicus Brevis): Week 148: number analyzed (Participants) | 10 | 36
  Right Abduction Thumb (Abductor Pollicus Brevis): Week 148 | -0.86 (1.861) | -1.10 (5.247)
  Right Abduction 5th Digit (Abductor Digiti Minimi): Week 52: number analyzed (Participants) | 25 | 41
  Right Abduction 5th Digit (Abductor Digiti Minimi): Week 52 | -0.78 (1.210) | -1.12 (5.112)
  Right Abduction 5th Digit (Abductor Digiti Minimi): Week 104: number analyzed (Participants) | 10 | 31
  Right Abduction 5th Digit (Abductor Digiti Minimi): Week 104 | -0.54 (1.059) | -0.21 (1.639)
  Right Abduction 5th Digit (Abductor Digiti Minimi): Week 148: number analyzed (Participants) | 10 | 36
  Right Abduction 5th Digit (Abductor Digiti Minimi): Week 148 | -0.69 (1.009) | -1.36 (5.634)
  Right Knee Extension: Week 52: number analyzed (Participants) | 25 | 42
  Right Knee Extension: Week 52 | -4.90 (5.964) | 1.05 (8.973)
  Right Knee Extension: Week 104: number analyzed (Participants) | 10 | 32
  Right Knee Extension: Week 104 | -2.16 (9.453) | -3.09 (13.046)
  Right Knee Extension: Week 148: number analyzed (Participants) | 10 | 35
  Right Knee Extension: Week 148 | -0.19 (7.407) | -1.60 (7.685)
  Right Ankle Dorsiflexion: Week 52: number analyzed (Participants) | 25 | 42
  Right Ankle Dorsiflexion: Week 52 | -5.68 (8.907) | -1.05 (5.923)
  Right Ankle Dorsiflexion: Week 104: number analyzed (Participants) | 10 | 32
  Right Ankle Dorsiflexion: Week 104 | -5.86 (3.501) | -3.78 (13.008)
  Right Ankle Dorsiflexion: Week 148: number analyzed (Participants) | 10 | 36
  Right Ankle Dorsiflexion: Week 148 | -6.74 (7.308) | -3.40 (8.172)

10. Secondary Outcome: 233AS101 and 233AS102 ISE: Time to Death or Permanent Ventilation
Description: Permanent ventilation was defined as ≥ 22 hours of mechanical ventilation [invasive or noninvasive] per day for ≥ 21 consecutive days. An event of permanent ventilation was based on an adjudicated event (i.e., adjudicated by the Endpoint Adjudication Committee (EAC) as having met the permanent ventilation criteria defined in the protocol). Time to death or permanent ventilation was defined as the time to the earliest occurrence of death or permanent ventilation. The start date for calculating time to death or permanent ventilation in days was date of first dose. Participants without an event were censored at the last known alive dates. This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on data collected from both 233AS101 & 233AS102 studies. This is reported as a part of final integrated analyses. Time to permanent ventilation or death was summarized using the Kaplan-Meier product limit method.
Time Frame: From the baseline of the study 233AS101 up to the end of the follow-up period of the current study (up to Week 364)
Population: Integrated analysis was performed on overall ITT population which included all Part C participants of 233AS101 and participants who rolled over from 233AS101 Part C into 233AS102. 'Overall number of participants analyzed' exceeds the total number of participants who started study 233AS102 as it indicates participants who were randomized in the Part C 233AS101 study.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
weeks | NA [135.6 to NA] — Due to the low number of events, the median and upper range of the 95% confidence interval (CI) were not estimable. | NA [253.6 to NA] — Due to the low number of events, the median and upper range of the 95% CI were not estimable.
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Test type: Superiority; p = 0.4202, Log Rank; The analysis was based on a log rank test stratified by median baseline plasma NfL; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.282 to 1.461] — The analysis was based on a Cox proportional hazards model adjusted for baseline plasma NfL, and riluzole or edaravone use

11. Secondary Outcome: 233AS101 and 233AS102 ISE: Time to Death
Description: Time to death was defined as the time from first dose received in 233AS101 to death. Participants who do not meet the endpoint definition were censored at the participant's last known alive date. Only events that were adjudicated by the EAC are included. This outcome measure was not a standalone analysis for 233AS102. Analysis was performed on data collected from both 233AS101 & 233AS102 studies. This is reported as a part of final integrated analyses. Time to death was summarized using the Kaplan-Meier product limit method.
Time Frame: From the baseline of the study 233AS101 up to the end of the follow-up period of the current study (up to Week 364)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg | 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg
Number analyzed (Participants) | 36 | 72
weeks | NA [NA to NA] — Due to the low number of events, the median and the 95% CI were not estimable. | NA [260.7 to NA] — Due to the low number of events, the median and upper range of the 95% CI were not estimable.
Statistical Analysis 1: Comparison: 233AS101 and 233AS102 (Part C): Placebo + Delayed-start BIIB067 100 mg vs 233AS101 and 233AS102 (Part C): Early-start BIIB067 100 mg; Test type: Superiority; p = 0.3108, Log Rank; The analysis was based on a log rank test stratified by median baseline plasma NfL; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.199 to 1.357] — [estimate comment as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of the study drug in the current study up to end of follow-up period (up to Week 364)
Description: The safety population included all participants who were enrolled and received at least one dose of study treatment in 233AS102.
Groups:
- 233AS101: Part C (Prior Placebo): Participants who were randomized to placebo in Part C of the parent study 233AS101 received 3 loading doses of BIIB067, 100 mg, Q2W, on Days 1, 15, and 29 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067, Q4W, until the last participant enrolled had their Week 152 maintenance dose visit.
- 233AS101: Part C (Prior BIIB067 100 mg): Participants who were randomized to BIIB067, 100 mg in Part C of the parent study 233AS101 received 2 loading doses of BIIB067, 100 mg on Days 1 and 29, and one dose of BIIB067-matched placebo on Day 15 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067, Q4W, until the last participant enrolled had their Week 152 maintenance dose visit.
- 233AS101: Parts A and B (All Doses): Participants who were randomized to BIIB067 in Part A (at doses 10 mg, 20 mg, 40 mg and 60 mg) or Part B (at doses 20 mg, 40, 60 mg and 100 mg) of the parent study 233AS101 received 3 loading doses of BIIB067, 100 mg, on Days 1, 15, and 29 by IT bolus injection in this study followed by up to 90 maintenance doses of BIIB067, Q4W, until the last enrolled participant had their Week 152 maintenance dose visit.
Arm/Group | 233AS101: Part C (Prior Placebo) | 233AS101: Part C (Prior BIIB067 100 mg) | 233AS101: Parts A and B (All Doses)
All-Cause Mortality (participants affected / at risk) | 7/32 | 14/63 | 5/44
Serious Adverse Events (participants affected / at risk) | 16/32 | 33/63 | 22/44
Other Adverse Events (participants affected / at risk) | 31/32 | 63/63 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 233AS101: Part C (Prior Placebo) (N=32) | 233AS101: Part C (Prior BIIB067 100 mg) (N=63) | 233AS101: Parts A and B (All Doses) (N=44)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 0
Myopericarditis (Cardiac disorders) | 0 | 0 | 1
Papilloedema (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 7 | 3
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 2 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 1
H1n1 influenza (Infections and infestations) | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Myelitis (Infections and infestations) | 1 | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1
Pneumonia aspiration (Infections and infestations) | 3 | 8 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 4
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 1
Brain hypoxia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1 | 0 | 0
Neurosarcoidosis (Nervous system disorders) | 0 | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 5
Euthanasia (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 233AS101: Part C (Prior Placebo) (N=32) | 233AS101: Part C (Prior BIIB067 100 mg) (N=63) | 233AS101: Parts A and B (All Doses) (N=44)
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 5
Conjunctivitis allergic (Eye disorders) | 2 | 0 | 0
Diplopia (Eye disorders) | 2 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 3
Papilloedema (Eye disorders) | 2 | 3 | 1
Vision blurred (Eye disorders) | 2 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 4
Constipation (Gastrointestinal disorders) | 10 | 12 | 11
Diarrhoea (Gastrointestinal disorders) | 12 | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 7 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 8 | 4
Nausea (Gastrointestinal disorders) | 7 | 13 | 17
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 13 | 2
Toothache (Gastrointestinal disorders) | 0 | 3 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3 | 7
Chills (General disorders) | 1 | 5 | 5
Fatigue (General disorders) | 10 | 16 | 13
Influenza like illness (General disorders) | 2 | 2 | 5
Malaise (General disorders) | 2 | 0 | 2
Oedema peripheral (General disorders) | 2 | 3 | 6
Pain (General disorders) | 3 | 5 | 2
Peripheral swelling (General disorders) | 2 | 3 | 5
Pyrexia (General disorders) | 8 | 11 | 11
Vaccination site pain (General disorders) | 0 | 4 | 1
Hepatic steatosis (Hepatobiliary disorders) | 3 | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 5 | 2
Bronchitis (Infections and infestations) | 1 | 3 | 6
Cellulitis (Infections and infestations) | 0 | 1 | 4
Covid-19 (Infections and infestations) | 7 | 26 | 13
Cystitis (Infections and infestations) | 3 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 3 | 4
Influenza (Infections and infestations) | 1 | 3 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 4
Nasopharyngitis (Infections and infestations) | 6 | 11 | 20
Oral candidiasis (Infections and infestations) | 2 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 4
Pneumonia (Infections and infestations) | 3 | 4 | 5
Pneumonia aspiration (Infections and infestations) | 2 | 3 | 0
Rhinitis (Infections and infestations) | 3 | 2 | 1
Sinusitis (Infections and infestations) | 4 | 4 | 3
Suspected covid-19 (Infections and infestations) | 2 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 7 | 9
Urinary tract infection (Infections and infestations) | 5 | 8 | 12
Viral infection (Infections and infestations) | 1 | 1 | 4
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 7 | 8 | 13
Fall (Injury, poisoning and procedural complications) | 18 | 25 | 28
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 4
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 2
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 2 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3 | 4
Muscle strain (Injury, poisoning and procedural complications) | 1 | 3 | 5
Neurological procedural complication (Injury, poisoning and procedural complications) | 2 | 4 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 6 | 15 | 13
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 3
Post procedural contusion (Injury, poisoning and procedural complications) | 3 | 2 | 2
Post procedural pruritus (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1 | 4
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 4 | 2
Procedural pain (Injury, poisoning and procedural complications) | 14 | 33 | 28
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 4 | 6
Skin laceration (Injury, poisoning and procedural complications) | 1 | 3 | 3
Traumatic lumbar puncture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Alanine aminotransferase increased (Investigations) | 2 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 2
Blood glucose increased (Investigations) | 1 | 2 | 4
Blood urine present (Investigations) | 0 | 2 | 4
Csf glucose increased (Investigations) | 0 | 4 | 2
Csf protein increased (Investigations) | 7 | 15 | 15
Csf white blood cell count increased (Investigations) | 2 | 15 | 11
Hepatic enzyme increased (Investigations) | 0 | 3 | 3
Oxygen saturation decreased (Investigations) | 2 | 1 | 0
White blood cell count increased (Investigations) | 0 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 19 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 27 | 26
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 11 | 11
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 10 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 7
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 14 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 17 | 19
Balance disorder (Nervous system disorders) | 2 | 2 | 4
Burning sensation (Nervous system disorders) | 1 | 1 | 3
Dizziness (Nervous system disorders) | 5 | 13 | 13
Dysarthria (Nervous system disorders) | 2 | 4 | 0
Headache (Nervous system disorders) | 17 | 35 | 31
Hypoaesthesia (Nervous system disorders) | 4 | 2 | 5
Intracranial pressure increased (Nervous system disorders) | 2 | 4 | 0
Migraine (Nervous system disorders) | 1 | 2 | 4
Muscle contractions involuntary (Nervous system disorders) | 2 | 6 | 4
Muscle spasticity (Nervous system disorders) | 2 | 3 | 2
Paraesthesia (Nervous system disorders) | 3 | 7 | 5
Pleocytosis (Nervous system disorders) | 3 | 5 | 7
Radicular pain (Nervous system disorders) | 1 | 0 | 3
Sciatica (Nervous system disorders) | 0 | 2 | 3
Sensory disturbance (Nervous system disorders) | 2 | 1 | 1
Tremor (Nervous system disorders) | 2 | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 6 | 3
Depression (Psychiatric disorders) | 0 | 5 | 5
Insomnia (Psychiatric disorders) | 3 | 6 | 5
Panic attack (Psychiatric disorders) | 0 | 1 | 3
Dysuria (Renal and urinary disorders) | 2 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 3 | 3 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 5
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 7
Hypotension (Vascular disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT03070119/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT03070119/SAP_001.pdf